CLINICAL TRIAL: NCT03592485
Title: Efficacy of Erector Spinae Plane Block and Pectoral Fascia Block in Patients Undergoing Mitral Valve Repair Through the Right Mini-thoracotomy
Brief Title: ESP vs ESP With PECS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Division of Cardiovascular Surgery, St. Jadwiga Provincial Clinical Hospital, Rzeszów, Poland (Unknown)
Responsible Party: Principal Investigator, Michał Borys, Principal Investigator, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/127/2018
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain; Mitral Valve Disease
Keywords: Erector Spinae Plane blockade; Pectoral Fascia block; patient control anlagesia; mitral valve replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Anesthesia, General; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP (Experimental): Before the induction of general anesthesia, Erector Spinae Plane (ESP) blockade will be done. Postoperative analgesia is provided with intravenous oxycodone. Patient-controlled analgesia pump (PCA) will be used for this purpose.
  Interventions: Procedure: Erector Spinae Plane blockade; Drug: Oxycodone; Procedure: general anesthesia; Drug: paracetamol
- PECS (Experimental): Before the induction of general anesthesia, Erector Spinae Plane (ESP) block and Pectoral fascia type I and II will be done. Postoperative analgesia is provided with intravenous oxycodone. Patient-controlled analgesia pump (PCA) will be used for this purpose.
  Interventions: Procedure: Erector Spinae Plane blockade; Procedure: Pectoral Fascia block; Drug: Oxycodone; Procedure: general anesthesia; Drug: paracetamol

INTERVENTIONS:
Procedure: Erector Spinae Plane blockade — Before the beginning of the procedure, ESP blockade will be performed under ultrasound control. A single-shot technique will be used with 0.375 % solution of ropivacaine: 0.1 mL per patients' KG. The maximum dose is 20 mL.
Procedure: Pectoral Fascia block — Before the beginning of the procedure, PECS type I and II blocks will be performed under ultrasound control. A single-shot technique will be used with 0.375 % solution of ropivacaine: 0.1 mL per patients' KG. The maximum dose is 20 mL.
  Arms: PECS
Drug: Oxycodone — Each patient, before the end of surgery, will be administered i.v. 0.1 mg of oxycodone. PCA with oxycodone (1mg/mL) will be utilized during the postoperative period: 5-minute interval.
Procedure: general anesthesia — Each patient will generally anesthetized and endotracheal tube will be inserted
  Other Names: GA
Drug: paracetamol — Paracetamol will be given i.v. every 6 hours.

SUMMARY:
Patients scheduled for minimally invasive mitral valve repair. Each patient will be treated with intravenous (i.v.) oxycodone - patient-controlled analgesia (PCA). Patients will be allocated to one of the groups: erector spinae plane (ESP) block or EPS with pectoral fascia (PECS) block.

DETAILED DESCRIPTION:
Only patients who are qualified for an elective procedure of mitral valve replacement may participate in the study. Each patient will be anesthetized generally. The same drugs will be used in each stage of anesthesia. The induction: etomidate, remifentanil, rocuronium, scolina as required. The maintenance: sevoflurane, remifentanil, rocuronium. The emergence: oxygen, sugammadex or neostigmine a required.

Patients will be randomly allocated to one of two groups: ESP or PECS. Among the patients from ESP group will have ESP blockade before the induction of general anesthesia. ESP blockade will be performed under ultrasound control. A single-shot technique will be used with 0.375 % solution of ropivacaine: 0.1 mL per patient KG. The maximum dose is 20 mL.

Patients from PECS group will receive ESP block and PECS I and II type block with 0.375 % solution of ropivacaine (up to 20 mL of local anesthetic).

Each patient, before the end of surgery, will be administered i.v. 0.1 mg of oxycodone. PCA with oxycodone (1mg/mL) will be utilized during the postoperative period: 7-minute interval. This is standard protocol in the investigator's department.

Only patients who are successfully awakened after the procedure may participate in the study.

The pain intensity will be assessed with visual-analogue scale (VAS) at 2, 4, 8, 12 and 24 hour after the end of anesthesia.

The total consumption of oxycodone will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled mitral valve replacement surgery
* obtained consent

Exclusion Criteria:

* allergy to oxycodone and local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs
* prolonged postoperative ventilation (over 2 hours)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Total consumption of oxycodone | From the end of anesthesia till 24 hour postoperatively
  The cumulative consumption of oxycodone during 24 hour from the end of anesthesia. Less is better, less intense pain.

SECONDARY OUTCOMES:
Pain intensity measured by VAS | From the end of anesthesia till 24 hour postoperatively
  Patient self-pain assessment on VAS (visual-analogue scale). VAS range from 0 (no pain, good outcome) to 100 in millimeters (the worst pain ever, bad outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiovascular Surgery, St. Jadwiga Provincial Clinical Hospital, Rzeszów, Poland, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaweda B, Borys M, Belina B, Bak J, Czuczwar M, Woloszczuk-Gebicka B, Kolowca M, Widenka K. Postoperative pain treatment with erector spinae plane block and pectoralis nerve blocks in patients undergoing mitral/tricuspid valve repair - a randomized controlled trial. BMC Anesthesiol. 2020 Feb 27;20(1):51. doi: 10.1186/s12871-020-00961-8. PMID 32106812